CLINICAL TRIAL: NCT01597154
Title: Beating Diabetes Together: A Randomized Controlled Trial for Intensive Lifestyle Therapy for Youth With Type 2 Diabetes
Brief Title: Lifestyle Therapy for Youth With Type 2 Diabetes
Acronym: BDT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Manitoba (Other)
Collaborators: Manitoba Institute of Child Health (Industry)
Responsible Party: Principal Investigator, Jon McGavock, Assistant Professor, University of Manitoba
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: B2012:023
Record Dates: First submitted 2012-05-09; First posted 2012-05-11 (Estimated); Last update posted 2014-07-29 (Estimated); Status verified 2014-07

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: Adolescent; Type 2 Diabetes; Peer mentorship
MeSH Terms: conditions — Diabetes Mellitus, Type 2

ARMS (2):
- Lifestyle counselling (Experimental): Exercise, nutrition and self-efficacy based lifestyle training in a peer mentoring setting
  Interventions: Behavioral: Lifestyle Counselling
- Control (No Intervention): Youth randomized to the control group will receive standard care for the first 16 weeks followed by 16 weeks of intervention

INTERVENTIONS:
Behavioral: Lifestyle Counselling — Participants will take part in 2-3 group based peer-led sessions per week in which they will learn about healthy lifestyle choices
  Arms: Lifestyle counselling

SUMMARY:
Background: Little is known about the efficacy of intensive lifestyle therapy (i.e. increased physical activity and dietary changes) for the management of glycemia and cardiometabolic risk factors in children and adolescents with type 2 diabetes (T2DM).

Our hypothesis is that education regarding healthy lifestyle changes will significantly reduce blood sugars in youth with T2DM that do not require insulin therapy. Our secondary hypothesis is that the intensive lifestyle therapy will cause quick and sustained reductions in health risk measured by body mass index (BMI), blood pressure, waist circumference, LDL cholesterol, serum triglycerides and apolipoprotein B.

DETAILED DESCRIPTION:
Youth between the ages of 10-20 years living with type 2 diabetes and not currently on insulin therapy will be randomly assigned to either a lifestyle intervention group or a control group. The lifestyle intervention group will meet 2-3 times per week for 16 weeks to take part in healthy living education sessions involving physical activity, healthy cooking, healthy gardening and how to start and sustain a healthy lifestyle change. At the beginning and end of the 16 weeks the investigators will measure the participants' blood sugars, height, weight, cholesterol, triglycerides and liver enzymes. The investigators will also take a picture of their kidney, heart and blood vessels using ultrasound. Those youth assigned to the control group will receive the 16 week intervention following their 16 week control period.

ELIGIBILITY:
Inclusion Criteria:

* youth with a BMI considered overweight according to the International Obesity Task Force
* diagnosed with type 2 diabetes, confirmed with a 2-hour oral glucose tolerance test within two years of enrollment

Exclusion Criteria:

* youth with type 1 diabetes
* use of insulin or other anti-diabetic drugs
* youth with medication-induced diabetes
* youth who have recently been admitted to hospital with ketoacidosis
* youth have experienced weight loss or enrolled in a weightloss program in the last 6 months
* youth with an orthapaedic injury preventing them from exercising
* youth who have a history of alcohol or drug abuse

Ages: 10 Years to 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 15 (Actual)
Dates: Start 2012-09; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Glycemic control determined by a standard fasting measure of glycosylated hemoglobin using internationally recognized DCCT assay | 16 weeks

SECONDARY OUTCOMES:
Cardiometabolic risk Z score | 16 weeks
  This is a composite score based on BMI z-score, waist circumference, c-reactive protein (CRP), fibrinogen, low density lipoprotein (LDL) and high density lipoprotein (HDL) cholesterol, triglycerides (TG) and apolipoprotein B (apoB), and a marker of fatty liver disease, alanine transaminase (ALT)
Presence of microalbuminuria | 16 weeks
  defined as a first morning albumin:creatinine ratio (ACR) 2.5-25 mg/mmol in a first morning urine collection
Hypertension | 16 weeks
  defined as a systolic blood pressure load >25% or a mean 24 hour systolic blood pressure >95th %ile for sex and height on 24 hour ambulatory blood pressure monitoring
Anthropometrics | 16 weeks
  Waist circumference in centimeters, body mass index (BMI) z-score and percent body fat will be assessed to determine if changes in body composition are associated with improvements in cardiometabolic risk
Cardiovascular structure and function | 16 weeks
  Vascular health will be assessed with non-invasive assessments of arterial stiffness, endothelium-dependant relaxation and carotid intima media thickness which will be treated as continuous variables. Left ventricular structure and function will be assessed using standard M-mode and doppler ultrasound techniques

CONTACTS AND LOCATIONS:
Overall Officials: Jonathon McGavock, PhD, Principal Investigator — University of Manitoba
Locations (1):
- Manitoba Institute of Child Health, Winnipeg, Manitoba, Canada